CLINICAL TRIAL: NCT00004150
Title: Pan-European Trials in Adjuvant Colon Cancer (PETACC-2): Randomized Phase III Intergroup Trial of High-Dose Infusional 5-FU (+ or - Folinic Acid) Versus Standard Bolus 5-FU/Folinic Acid
Brief Title: High-Dose Fluorouracil With or Without Leucovorin Compared With Standard Fluorouracil Plus Leucovorin Following Surgery in Treating Patients With Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert Roessle Klinik (Individual)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Federation Francophone de Cancerologie Digestive (Other); Grupo Espanol Tratamiento Tumores Digestivos (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067383; PETACC-2; EORTC-40963; FFCD-PETACC-2; GETTD-PETACC-2
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2001-02

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; adenocarcinoma of the colon; mucinous adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which chemotherapy regimen is more effective for colon cancer.

PURPOSE: This randomized phase III trial is studying high-dose fluorouracil with or without leucovorin to see how well it works compared to standard-dose fluorouracil and leucovorin in treating patients who have undergone surgery for stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare recurrence-free survival and duration of survival in patients with stage III adenocarcinoma of the colon treated with adjuvant high-dose fluorouracil with or without leucovorin calcium versus standard fluorouracil with leucovorin calcium following curative radical resection.
* Compare the safety of these regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to regional lymph node involvement (N1 (1-3 pericolic lymph nodes) vs N2 (more than 3 pericolic lymph nodes) and participating center.

Patients are randomized to one of two treatment arms.

* Arm I: Patients receive leucovorin calcium IV followed by fluorouracil IV on days 1-5. Treatment repeats every 4 weeks for 6 courses.
* Arm II: Patients receive high-dose fluorouracil IV continuously over 48 hours weekly for 8 weeks. Treatment repeats every 8 weeks for 3 courses.

OR

* Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 24 hours weekly for 6 weeks. Treatment repeats every 7 weeks for 3 courses.

OR

* Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV bolus and then fluorouracil IV continuously over 22 hours on days 1 and 2. Treatment repeats every 2 weeks for 12 courses.

Patients are followed at 1 month, every 6 months for 4.5 years, and then annually thereafter until death.

PROJECTED ACCRUAL: Approximately 1,600 patients (800 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III adenocarcinoma or mucinous adenocarcinoma of the colon
* Must have had curative radical resection within 56 days prior to study

  * No local tumor therapy (i.e., polypectomy, local excision or limited intestinal resection)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No severe coronary heart disease
* No New York Heart Association class III or IV heart failure

Other:

* No other malignancy within the past 10 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled infection
* No other severe disease
* No known allergy to leucovorin calcium
* No known familial adenomatous polyposis, Crohn's disease, or ulcerative colitis
* No hereditary syndrome (e.g., Gardner's syndrome, Turcot's syndrome, hereditary nonpolyposis colon cancer)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for colon cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for colon cancer

Surgery:

* See Disease Characteristics

Other:

* No other concurrent systemic anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus-Henning Koehne, MD — Klinikum Oldenburg; G. Leam — Saint Laurentius Ziekenhuis; Laurent Bedenne, MD — Hopital Du Bocage; Alfredo Carrato-Mena, MD, Study Chair — Hospital Universitario de Elche
Locations (85):
- Belgium (7):
  - Ziekenhuis Network Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- France (39):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Clinique St. Etienne, Bayonne
  - Centre Hospitalier General, Belfort
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Clinique du Cedre, Bois-Guillaume
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier de Bourgoin - Jallieu, Bourgoin
  - Centre Hospitalier General, Brivé
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier de Chalons - en - Champagne, Châlons-en-Champagne
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Clinique Pasteur, Évreux
  - Cabinet de Gastro-Enterologie, Les Sables-d'Olonne
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Hopital de la Croix Rousse, Lyon
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Clinique du Pont de Chaume, Montauban
  - Hopital St. Eloi, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hopital de l'Archet, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Cochin, Paris
  - Clinique Ste - Marie, Pontoise
  - Institut Jean Godinot, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Hospitalier D'Agen, Saint-Esprit
  - Centre Hospitalier General de Saint Nazaire, Saint-Nazaire
  - Centre Paul Strauss, Strasbourg
  - CHU Rangueil, Toulouse
  - Nouvelle Clinique Generale, Valence
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier General - St. Nicolas, Verdun
  - Centre Hospitalier Regionale de Vichy, Vichy
  - Institut Gustave Roussy, Villejuif
- Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin, Germany
- Saint Laurentius Ziekenhuis, Roermond, Netherlands
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Spain (36):
  - Hospital General, Albacete
  - Hospital Virgen de los Lirios, Alcoi Alicante
  - Hospital General - Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de Barbastro, Barbastro
  - Hospital Del Mar, Barcelona
  - Institut d'Oncologia Corachan, Barcelona
  - Hospital de la Santa Cruz I Sant Pau, Barcelona
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Consorci Hospitalari de la Creu Roia, Barcelona
  - Hospital de L'esperit Sant, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Universarito "Reina Sofia", Córdoba
  - Hospital Virgen de Luz, Cuenca
  - Hospital Universitario de Elche, Elche Alicante
  - Hospital General Virgen de las Nieves, Granada
  - Hospital General Universitario De Guadalajara, Guadalajara
  - Residencia Sanitaria de Jaen, Jaén
  - Hospital General de Jerez, Jerez de la Frontera
  - Fundacion Jimenez Diaz - Clin. N.S., Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Regional Carlos Haya De Malaga, Málaga
  - Hospital De Merida, Mérida
  - Hospital De Navarra, Pamplona
  - Consorci Hospitalari del Parc Tauli, Sabadell
  - Hospital de Sagunto, Sagunto
  - Hospital Virgen de la Vega, Salamanca
  - Hospital Universitario Canarias, San Cristóbal de La Laguna
  - Hospital Universitari Sant Joan d'Alacant, San Juan
  - Hospital - Residencia Sant Camil, Sant Pere de Ribes
  - Hospital Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife
  - Hospital Consorci Sanitari De Terrassa, Terrassa
  - Instituto Valenciano De Oncologia, Valencia
  - Hospital General Universitario Valencia, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Fensterer H, Radlwimmer B, Strater J, Buchholz M, Aust DE, Julie C, Radvanyi F, Nordlinger B, Belluco C, Van Cutsem E, Kohne CH, Kestler HA, Schwaenen C, Nessling M, Lutz MP, Lichter P, Gress TM; EORTC Gastrointestinal (GI) Group. Matrix-comparative genomic hybridization from multicenter formalin-fixed paraffin-embedded colorectal cancer tissue blocks. BMC Cancer. 2007 Apr 2;7:58. doi: 10.1186/1471-2407-7-58. PMID 17407575
- [Result] Carrato A, Köhne C, Bedenne L, et al.: Folinic acid modulated bolus 5-FU or infusional 5-FU for adjuvant treatment of patients of UICC stage III colon cancer: preliminary analysis of the PETACC-2-study. [Abstract] J Clin Oncol 24 (Suppl 18): A-3563, 2006.